CLINICAL TRIAL: NCT02497989
Title: Male Circumcision for HIV Prevention in Kenya: Seeking Effective Strategies to Recruit Older Men
Brief Title: Evaluating Demand Creation Strategies for Voluntary Medical Male Circumcision (VMMC) in Kenya
Acronym: TASCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Impact Research & Development Organization (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Kenya Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Kawango Agot, Director, Impact Research & Development Organization
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: GH000518
Record Dates: First submitted 2015-05-20; First posted 2015-07-15 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: HIV/AIDS
Keywords: Male circumcision; Demand creation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Inter-personal Communication (IPC) (Experimental): Interpersonal communication will entail delivery of intervention massages that are custom-made to address individual participants' specific barriers and facilitators of VMMC. RAs will discuss with uncircumcised men why they have not gone for VMMC using the 'VMMC Demand Creation Toolkit'. The aim will be to fully address their barriers and re-enforce their facilitators. RAS will be trained behavioral counselors, circumcised men, female partners, CHWs, or any other cadre of individuals identified during the formative phase.
  Interventions: Other: Inter-personal Communication (IPC)
- Dedicated Service Outlets (DSO) (Experimental): RAs shall visit all households with eligible men to inform them about the availability of, and give information on location of DSO sites in the Location. DSOs are sites: where services are offered exclusively to men aged ≥25 years by male service providers in the same age bracket; providing services in the evenings/weekends/designated days of the week, and through special mobile services for older men. DSO sites we will strive to shorten the waiting time to ≤ three hours. They will be informed that all other VMMC sites continue to serve all men regardless of age (i.e., including older men) while DSO sites will only serve men aged ≥25 years. RAs will respond to questions using 'All You Need to Know About VMMC' booklet, the same way current recruiters do.
  Interventions: Other: Dedicated Service Outlets (DSO)
- Combined IPC & DSO (Experimental): Both Inter-personal Communication (IPC) and Dedicated Service Outlets (DSO) interventions (as described above) will be implemented concurrently. This will be done to determine the effect of both interventions delivered jointly compared to each delivered singly, and compared to no intervention.
  Interventions: Other: Inter-personal Communication (IPC); Other: Dedicated Service Outlets (DSO)
- Control (No Intervention): In these Locations, participants will only be given the 'All You Need to Know About VMMC' booklet at the time of enrollment, which is the standard of care.

INTERVENTIONS:
Other: Inter-personal Communication (IPC) — RAs will meet older men in their households, and : i) approach the person(s), introduce self, develop rapport and request for time to discuss briefly about VMMC; ii) strike a conversation on reasons why they or their peers have not gone to be circumcised as well as reasons that would make them get circumcised, jotting down responses to guide the discussion; iii) using the 'VMMC Demand Creation Toolkit', discuss each reported barrier/facilitator carefully and completely, always ensuring the person(s) is/are engaged in the discussion (the goal is to pass correct and complete information in a relaxed and conversational manner); iv) revisiting each stated barrier/barrier and exploring what they now think about them after the discussion, and address any new or lingering concerns.
  Arms: Combined IPC & DSO; Inter-personal Communication (IPC)
Other: Dedicated Service Outlets (DSO) — RAs shall visit every household with eligible men to inform them about the availability of DSO sites in their neighborhoods. After describing the characteristics of DSO sites, the RA will share - both verbally and through a flyer, information on where to find DSO sites in the respective Location. RAs will respond to questions using 'All You Need to Know About VMMC' booklet, the same way current recruiters do. They will also inform potential participants that all other VMMC sites continue to serve all men regardless of age (i.e., including older men) while DSO sites will only serve men aged ≥25 years.
  Arms: Combined IPC & DSO; Dedicated Service Outlets (DSO)

SUMMARY:
The purpose of this study is to evaluate the impact of two interventions - Inter-Personal Communication [IPC] and Dedicated Service Outlets [DSOs] - in recruiting men aged 25-39 years for Voluntary Medical Male Circumcision (VMMC) services.

DETAILED DESCRIPTION:
STUDY AIMS Aim 1: Assess the rate of uptake of VMMC services by men aged 25-39 years exposed to Inter-Personal Communication (IPC) vs. Designated (older men only) Service Outlets (DSO) vs. IPC and DSO interventions combined vs. no intervention.

Aim 2: Determine through testing of unlinked de-identified blood from bleeding vessels from the surgical wound, the proportion of men whose HIV status is unknown who are HIV infected (Sub-study 1).

Aim 3: Determine the cost of providing VMMC among the three interventions relative to each other and to no intervention.

MAIN STUDY DESIGN: The study proposes to conduct a cluster randomized-controlled trial, with Locations forming the unit of randomization. Within the selected Locations, the study shall randomly select approximately 16% (209) of the villages which will be sufficient to generate the required sample size.

Sample size Determination:

Sample size for detecting the impact of the interventions on VMMC uptake - in order to be able demonstrate at least a 33.3 % increase in the rate of VMMC among young adult men in intervention arms when compared to those in control arm with 80% statistical power, and Bonferroni adjusted two-sided α=(0.05/3)=0.017 following the implementation of study interventions, the study will need a sample size of 4,932 men reached with the intervention.

Potential participants to be reached - An effect size equal to 33.3% increase in MC from 30% to 40% will require about 1233 participants per study arm (total 4932), while an effect size equal to 50% increase in VMMC from 30% to 45% will require 573 participants per study arm (total 2292). Adjusting for a refusal rate of 15% and a loss to follow up of 15%, suggests contacting 1603 per study arm resulting in a total of 6412 uncircumcised men aged 25-39 years.

PHASE 1: HOUSEHOLD ENUMERATION To ascertain the size of eligible population (uncircumcised men aged 25-39 years), the study will conduct complete household listing in all selected villages and enumerate male members in each household aged 25-39 years. During this exercise, study staff shall physically visit all homes in the study villages and assign a unique identification number to every household (HIN). Enumeration shall be through home visits ONLY and not by any other means. The unique HIN assigned during the enumeration will be entered on Excel database and households with men aged 25-39 years will be sorted out and put on a separate list. The list will be used to create a database of eligible men in each village. Determining the number of households with eligible men will help in knowing the denominator and in planning for recruitment.

PHASE 2: CONDUCTING RAPID FORMATIVE STUDY (Sub-study 1) Justification: This phase is intended to provide information for use in delivering the interventions. The study have already drafted messages based on existing literature for use in IPC and IPC+DSO intervention Locations/villages. However, since almost all the available information on barriers to and facilitators of VMMC in literature were collected among men of all ages and were not disaggregated by age group, the investigators cannot assume they are automatically relevant to older men. As such, it will still be necessary to conduct a rapid formative study to explore reasons why older men aged 25-39 years go or do not go for VMMC services. Information obtained from this phase will be used to modify if indicated, the messages developed from existing literature.

SUB-STUDY DESIGN: This phase shall comprise of Focus Group Discussions (FGDs) and In-Depth Interviews. Twelve FGDs, with 6-10 participants, will be held with six groups of circumcised men and six groups of uncircumcised men in each of the following age categories: 25-29 years, 30-34 years and 35-39 years. A similar number of FGDs will be held with female partners of circumcised and female partners of uncircumcised men in same age categories.

Besides FGDs, the investigators will conduct 48 IDIs to capture confidential information that some men and women would otherwise not divulge in an FGD setting.

PHASE 3: ESTABLISHING BASELINE VMMC PREVALENCE AND PROPORTION OF ELIGIBLE MEN Based on the eligible participants' list, research assistants will only go back to households with men aged 25 to 39 years. Before administering enrollment consent, RAs will ask participants to identify a private location within or outside the house where they can do consenting and interviewing. The RA will then administer consent for participating in the study, enrol consenting participants and assign Participant Unique ID number.

After assigning the participant unique ID number, the RA will conduct the baseline interview, verify the MC status and inform participants of their intervention arm and deliver the intervention if the participant is available (if not, another visit will be made at a later date to deliver the intervention). During the interview, study staff will document participants' circumcision status from the verbal report. After the interview, participants who consented to physical verification will be asked to choose where this can be performed.

At enrollment, participants will be given 3 months within which to go for circumcision, Participants can go whenever they want for VMMC, but the study will only capture their data if they go within 3 months. They will also be informed that a reminder of the expiry date for circumcision will be sent through text message to all participants one month before the expiry of the circumcision window period.

Details of participants enrolled in the study will be entered into an excel Master Log which will contain all participant details; 3 names, ID number, age, location, village, the telephone number of the participants or of close friend and date of enrollment.

PHASE 4: IMPLEMENTING THE INTERVENTIONS The study has four intervention arms: Inter-Personal Communications (IPC), Dedicated Service Outlets (DSOs), a combination of IPC and DSO (IPC+DSO), and Control. The interventions and how each of them will be implemented are described under 'Protocol arms and interventions' section below.

HIV TESTING OF PARTICIPANTS WITH UNKNOWN HIV STATUS (Sub-study 2) In VMMC program undertaken by Impact Research and Development Organization (IRDO) and in other Kenyan programs as well, between 10% and 30% of men decline HIV testing. Given that VMMC is offered principally as an HIV prevention strategy, it is important to determine the HIV status of those who decline testing, and if the prevalence is significantly higher than those who accept testing, there will be need to design approaches to improve uptake of testing. This is particularly important following results from a recently concluded study that indicated that 44% of HIV-infected men resumed sex before the recommended 6 weeks of sexual abstinence.

Sample size for HIV prevalence among uncircumcised men whose HIV status is unknown (Sub-study 2):

Investigators estimated that they will need to test randomly selected unlinked blood samples from 163 men per arm whose HIV status is unknown in order to estimate a HIV prevalence that falls within 10% points of the true population prevalence with 95% confidence. The study staff will collect samples from all of men who refuse testing but consent to Unlinked HIV testing.

With a refusal rate of 23.6% voluntary HIV testing, and a consenting rate of 60%, then the rate of getting a man who refuses testing but consents to the testing of unlinked blood sample from his bleeding vessels is 14.2%. In other words, of the 4932 participants in the main study, investigators expect 1164 (4932*0.236) to refuse HIV testing. With assumed unlinked HIV testing acceptance rate of 60%, the study can obtain 700 such men from a sample size of 4932 in the main study. For a design effect of 2.5, using a sample size of 700 for the sub-study will enable us to estimate the HIV prevalence of 21.6% with a precision of 4.8%=sqrt[(2.5*1.96^2*.216*.784)/700].

Methods/Procedure:

RAs will perform unlinked testing of blood from bleeding vessels or finger prick of those whose HIV status is unknown. While the call for proposals recommended testing blood from the excised foreskin, investigators are concerned that they may not be able to harvest sufficient blood from most foreskins to perform the test. This is because the forceps-guided method being used in Kenya crushes the foreskin and compresses the blood vessels that supply the distal section. This results in little or no bleeding on the excised foreskin. The study, therefore, propose to only collect blood samples from the bleeding vessels or finger prick from participants (n=700).

COSTING VMMC IN THE CONTEXT OF THE INTERVENTIONS (SUB-STUDY 3) Study Design: Data on costing will be collected across all the study arms. Whereas economic evaluation of service delivery has been conducted in several contexts there is limited information on the cost-effectiveness of various approaches used for recruitment to increase service uptake. The study plan to assess the cost-effectiveness of demand creation for VMMC services based on the three interventions. The results will demonstrate the accrued costs and net savings associated with each intervention strategy.

Methods: The primary outcome of the main study is the incremental change in circumcisions performed attributable to the respective demand creation interventions. Costs will be estimated for primary outcome with reference to the control group, in which the study will continue to provide routine recruitment approaches. This will demonstrate how the costs vary depending on the mode of demand creation.

The study shall adopt a societal perspective because of the ability to integrate diverse factors into the model and the role the public sector plays in HIV prevention and management. This approach incorporates all costs borne by the implementers in recruiting participants for services.

Sources of costing data:

The study will collect data from all study sites using a tool adapted from the Male Circumcision Decision-Makers' Program Planning Tool (DMPPT) for each of the demand creation strategies. The DMPPT was developed by the USAID/Health Policy Initiative in collaboration with UNAIDS to enable decision-makers to understand the potential cost and impact of various options for scaling up male circumcision services. The DMPPT has previously been used to undertake costing of male circumcision services in East and Central Africa. The study shall use this instrument as a data collection tool to estimate the cost of demand creation and the unit cost of providing VMMC (i.e. cost per adult circumcised) in each of the four study arms.

PHASE 5: ESTABLISHING ENDLINE MC PREVALENCE/ESTIMATING IMPACT OF INTERVENTIONS At Endline, the study will review Participant Master Log to identify those who did not go for VMMC at the 45 VMMC clinics participating in the study. The study will use the telephone numbers obtained during enrollment to contact the participants. Those who say that they got circumcised but are not in the Participant Master Log, study staff will make an appointment and visit them at home, or another convenient location, to administer consent, conduct Endline interview and verify their circumcision status. Those who report not having gone for VMMC will be asked why they did not go, and their response recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Uncircumcised men
2. Aged 25 - 39 years
3. Residents of the study village (has been living in the physical structure such as a compound or homestead identified during the enumeration and who has been consuming or making some contribution to food and other shared household resources).
4. Intend to continue living in the village for the 9 months after enrollment, which is the estimated duration of data collection.
5. Give written consent to participate in the study and the interventions.

Exclusion Criteria:

1. Circumcised men
2. Aged <25- or >39 years
3. Non-resident of target villages
4. Plans to move away from the village within 9 months after enrollment
5. Does not give consent to participate in the study

Ages: 25 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2785 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01-22 (Actual)

PRIMARY OUTCOMES:
The rate of uptake of VMMC services among men in 4 study arms | Three months post intervention
  We will assess the rate of uptake of VMMC services by men aged 25-39 years exposed to (i) Inter-personal communication (IPC) intervention vs. (ii) Designated (older men only) Service Outlets (DSO) intervention vs. (iii) IPC and DSO interventions combined vs. (iv) No intervention.

SECONDARY OUTCOMES:
Prevalence of HIV among VMMC clients who decline HIV testing | Three months post intervention
  Determine HIV prevalence among men in the study target group who refuse routine HIV testing but consent to the testing of unlinked blood sample from bleeding vessels or finger prick.

OTHER OUTCOMES:
Cost of VMMC demand creation | Nine months
  Determine the overall cost of VMMC demand creation, as well as the unit cost of providing VMMC services under each of the proposed 3 demand creation strategies.
Role of female sexual partners in time to resumption of sex post circumcision | Nine months
  The level of involvement of female sexual partners in their partners' decisions and activities before, during and after circumcision and the association between the level of partner involvement in circumcision decision-making and the length of post-surgical sexual abstinence, condom use, and sexual partnerships.

CONTACTS AND LOCATIONS:
Overall Officials: Kawango Agot, PhD, MPH, Principal Investigator — Impact Research and Development Organization; Jonathan Grund, MA, MPH, Principal Investigator — Centers for Disease Control and Prevention; Jacob Onyango, Study Director — Impact Research and Development Organization
Locations (1):
- Impact Research and Development Organization, Kisumu, Nyanza, Kenya

REFERENCES:
- [Background] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Background] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Weiss HA, Halperin D, Bailey RC, Hayes RJ, Schmid G, Hankins CA. Male circumcision for HIV prevention: from evidence to action? AIDS. 2008 Mar 12;22(5):567-74. doi: 10.1097/QAD.0b013e3282f3f406. No abstract available. PMID 18316997
- [Background] Siegfried N, Muller M, Deeks JJ, Volmink J. Male circumcision for prevention of heterosexual acquisition of HIV in men. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD003362. doi: 10.1002/14651858.CD003362.pub2. PMID 19370585
- [Background] UNAIDS/WHO/SACEMA Expert Group on Modelling the Impact and Cost of Male Circumcision for HIV Prevention. Male circumcision for HIV prevention in high HIV prevalence settings: what can mathematical modelling contribute to informed decision making? PLoS Med. 2009 Sep;6(9):e1000109. doi: 10.1371/journal.pmed.1000109. Epub 2009 Sep 8. PMID 19901974
- [Background] Weiss HA, Quigley MA, Hayes RJ. Male circumcision and risk of HIV infection in sub-Saharan Africa: a systematic review and meta-analysis. AIDS. 2000 Oct 20;14(15):2361-70. doi: 10.1097/00002030-200010200-00018. PMID 11089625
- [Background] Nagelkerke NJ, Moses S, de Vlas SJ, Bailey RC. Modelling the public health impact of male circumcision for HIV prevention in high prevalence areas in Africa. BMC Infect Dis. 2007 Mar 13;7:16. doi: 10.1186/1471-2334-7-16. PMID 17355625
- [Background] Njeuhmeli E, Forsythe S, Reed J, Opuni M, Bollinger L, Heard N, Castor D, Stover J, Farley T, Menon V, Hankins C. Voluntary medical male circumcision: modeling the impact and cost of expanding male circumcision for HIV prevention in eastern and southern Africa. PLoS Med. 2011 Nov;8(11):e1001132. doi: 10.1371/journal.pmed.1001132. Epub 2011 Nov 29. PMID 22140367
- [Background] Bailey RC, Egesah O, Rosenberg S. Male circumcision for HIV prevention: a prospective study of complications in clinical and traditional settings in Bungoma, Kenya. Bull World Health Organ. 2008 Sep;86(9):669-77. doi: 10.2471/blt.08.051482. PMID 18797642
- [Background] Rennie S, Muula AS, Westreich D. Male circumcision and HIV prevention: ethical, medical and public health tradeoffs in low-income countries. J Med Ethics. 2007 Jun;33(6):357-61. doi: 10.1136/jme.2006.019901. PMID 17526688
- [Background] Herman-Roloff A, Otieno N, Agot K, Ndinya-Achola J, Bailey RC. Acceptability of medical male circumcision among uncircumcised men in Kenya one year after the launch of the national male circumcision program. PLoS One. 2011;6(5):e19814. doi: 10.1371/journal.pone.0019814. Epub 2011 May 16. PMID 21603622
- [Background] Ngalande RC, Levy J, Kapondo CP, Bailey RC. Acceptability of male circumcision for prevention of HIV infection in Malawi. AIDS Behav. 2006 Jul;10(4):377-85. doi: 10.1007/s10461-006-9076-8. PMID 16736112
- [Background] Ivers NM, Taljaard M, Dixon S, Bennett C, McRae A, Taleban J, Skea Z, Brehaut JC, Boruch RF, Eccles MP, Grimshaw JM, Weijer C, Zwarenstein M, Donner A. Impact of CONSORT extension for cluster randomised trials on quality of reporting and study methodology: review of random sample of 300 trials, 2000-8. BMJ. 2011 Sep 26;343:d5886. doi: 10.1136/bmj.d5886. PMID 21948873
- [Background] Marya Plotkin, Hawa Mziray, Jan Küver Judith Prince, et al (2011). Embe Halijamenywa: The unpeeled mango: A Qualitative Assessment of Views and Preferences concerning Voluntary Voluntary Medical Male Circumcision in Iringa Region, Tanzania.
- [Background] KNBS (2010) 2009 Kenya Population and Housing Census, Volume I A; Population by Administrative Units, Kenya National Bureau of Statistics, Nairobi, Kenya
- [Background] E.Odoyo-June , J H Rogers, W Jaoko, et al. Sex before wound healing and condom use among newly circumcised HIV-positive and HIV-negative men in Kisumu, Kenya. 19th International AIDS Conference. Abstract no MOPE170
- [Background] Czarnogorski M, Brown J, Lee V, Oben J, Kuo I, Stern R, Simon G. The Prevalence of Undiagnosed HIV Infection in Those Who Decline HIV Screening in an Urban Emergency Department. AIDS Res Treat. 2011;2011:879065. doi: 10.1155/2011/879065. Epub 2011 May 9. PMID 21738860
- [Background] Weinstock H, Dale M, Linley L, Gwinn M. Unrecognized HIV infection among patients attending sexually transmitted disease clinics. Am J Public Health. 2002 Feb;92(2):280-3. doi: 10.2105/ajph.92.2.280. PMID 11818306
- [Background] Dukers-Muijrers NH, Niekamp AM, Vergoossen MM, Hoebe CJ. Effectiveness of an opting-out strategy for HIV testing: evaluation of 4 years of standard HIV testing in a STI clinic. Sex Transm Infect. 2009 Jun;85(3):226-30. doi: 10.1136/sti.2008.033191. Epub 2008 Dec 22. PMID 19103641
- [Background] National AIDS and STI Control Programme NASCOP (2008). Adapted by the Male Circumcision Task Force, Ministry of Health, Kenya, from the WHO/UNAIDS/JHPIEGO Manual for Male Circumcision under Local Anaesthesia. Version 2.5C, February 2008.
- [Background] Bertrand JT, Njeuhmeli E, Forsythe S, Mattison SK, Mahler H, Hankins CA. Voluntary medical male circumcision: a qualitative study exploring the challenges of costing demand creation in eastern and southern Africa. PLoS One. 2011;6(11):e27562. doi: 10.1371/journal.pone.0027562. Epub 2011 Nov 29. PMID 22140450
- [Background] Bollinger L W, Plosky D, Stover J. (2009). Male circumcision: Decision Maker's Program Planning Tool, calculating the costs and Impacts of a Male Circumcision Program. Washington, DC: Futures Group, Health Policy Initiative , Task Order 1
- [Background] Kahn JG, Marseille E, Auvert B. Cost-effectiveness of male circumcision for HIV prevention in a South African setting. PLoS Med. 2006 Dec;3(12):e517. doi: 10.1371/journal.pmed.0030517. PMID 17194197
- [Background] Schroeder E, Petrou S, Patel N, Hollowell J, Puddicombe D, Redshaw M, Brocklehurst P; Birthplace in England Collaborative Group. Cost effectiveness of alternative planned places of birth in woman at low risk of complications: evidence from the Birthplace in England national prospective cohort study. BMJ. 2012 Apr 18;344:e2292. doi: 10.1136/bmj.e2292. PMID 22517916
- [Background] Gray RH, Li X, Kigozi G, Serwadda D, Nalugoda F, Watya S, Reynolds SJ, Wawer M. The impact of male circumcision on HIV incidence and cost per infection prevented: a stochastic simulation model from Rakai, Uganda. AIDS. 2007 Apr 23;21(7):845-50. doi: 10.1097/QAD.0b013e3280187544. PMID 17415039
- [Background] Tekeste A, Wondafrash M, Azene G, Deribe K. Cost effectiveness of community-based and in-patient therapeutic feeding programs to treat severe acute malnutrition in Ethiopia. Cost Eff Resour Alloc. 2012 Mar 19;10:4. doi: 10.1186/1478-7547-10-4. PMID 22429892
- [Background] Prinja S, Bahuguna P, Rudra S, Gupta I, Kaur M, Mehendale SM, Chatterjee S, Panda S, Kumar R. Cost effectiveness of targeted HIV prevention interventions for female sex workers in India. Sex Transm Infect. 2011 Jun;87(4):354-61. doi: 10.1136/sti.2010.047829. Epub 2011 Mar 29. PMID 21447514
- [Background] Evans DB, Edejer TT, Adam T, Lim SS. Methods to assess the costs and health effects of interventions for improving health in developing countries. BMJ. 2005 Nov 12;331(7525):1137-40. doi: 10.1136/bmj.331.7525.1137. No abstract available. PMID 16282411
- [Background] Ioannidis JP, Garber AM. Individualized cost-effectiveness analysis. PLoS Med. 2011 Jul;8(7):e1001058. doi: 10.1371/journal.pmed.1001058. Epub 2011 Jul 12. PMID 21765810
- [Background] National AIDS Control Council 2. (NACC), N.A.C.C., The Kenya National HIV/AIDS Strategic Plan 2010-2013 (KNASP III). 2009: Nairobi, Kenya.. (2009). The Kenya National HIV/AIDS Strategic Plan 2010 - 2013 (KNASP III). Ministry of Public Health and Sanitation, Nairobi, Kenya.
- [Background] Male Circumcision Consortium 1. (MCC), M.C.C. 2011. News. December 2011; issue 33
- [Derived] Grund JM, Onchiri F, Mboya E, Ussery F, Musingila P, Ohaga S, Odoyo-June E, Bock N, Ayieko B, Agot K. Strategies to increase uptake of voluntary medical male circumcision among men aged 25-39 years in Nyanza Region, Kenya: Results from a cluster randomized controlled trial (the TASCO study). PLoS One. 2023 Feb 3;18(2):e0276593. doi: 10.1371/journal.pone.0276593. eCollection 2023. PMID 36735665